CLINICAL TRIAL: NCT03292497
Title: Prospective Treatment Algorithm Guiding Repair of Severe Ischemic Mitral Regurgitation: Canadian Mitral Research Alliance (CAMRA) 2 Trial
Brief Title: Prospective Treatment Algorithm Guiding Repair of Severe Ischemic Mitral Regurgitation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20170700
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Echocardiographic outcome assessment will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment algorithm (Experimental): Mitral valve will be replaced if posterior leaflet tethering angle >=25 degrees.
  Mitral valve will be repaired if posterior leaflet tethering angle <25 degrees
  Interventions: Procedure: Treatment Algorithm
- No treatment algorithm (Active Comparator): Mitral valve will be repaired or replaced at surgeon's discretion.
  Interventions: Procedure: No Treatment Algorithm

INTERVENTIONS:
Procedure: Treatment Algorithm — Patients will have their procedure dictated by a treatment algorithm. They will have their mitral valve replaced if the posterior leaflet tethering angle >=25 degrees, or repaired if the posterior leaflet tethering angle <25 degrees.
  Arms: Treatment algorithm
Procedure: No Treatment Algorithm — Patients will have their valve repaired or replaced at the discretion of their surgeon.
  Arms: No treatment algorithm

SUMMARY:
Ischemic mitral regurgitation is a disease where the mitral valve is regurgitant, or leaking, as a result of changes in the muscle of the heart caused by coronary artery disease Ischemic mitral regurgitation, or IMR, is normally treated by repairing or replacing the mitral valve. Currently, we don't have very strong evidence showing which patients might benefit from mitral valve repair and which might benefit from replacement, and surgeons tend to repair or replace valves based on their preference or experience. Some surgeons, including Dr. Vincent Chan, the Principal Investigator, believe that the decision to repair or replace the valve should be based on specific measurements of the mitral valve. This study will randomly assign patients to receive either the current standard of care for ischemic mitral regurgitation, which is valve repair or replacement based on the surgeon's preference, or to have their treatment decided by a set of criteria called an algorithm. This algorithm will assign patients with certain mitral valve measurements to repair, and others to replacement. Patients will be followed for 12 months after surgery, to compare whether patients whose treatment was decided by the algorithm did better than patients whose treatment was decided by surgeon preference.

ELIGIBILITY:
Inclusion Criteria:

* Severe ischemic mitral valve regurgitation

  * 18 years of age, and able to provide informed consent.

Exclusion Criteria:

* Mixed mitral valve pathology
* Acute ischemic mitral regurgitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2018-01-16 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Left ventricle end-systolic volume indexed to body surface area | 12 months after surgery
  Comparison of changes in the indexed volume of the left ventricle.

SECONDARY OUTCOMES:
Change in indexed left atrial volume | Up to 12 months after surgery
  Comparison of changes in the indexed volume of the left atrium.
Change in right ventricle systolic pressure | Up to 12 months after surgery
  Comparison of changes in the systolic pressure of the right ventricle.
Major adverse events | Up to 12 months after surgery
  Composite endpoint of survival, recurrence of clinically-significant (>= 2+) mitral regurgitation, and readmission to hospital for congestive heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Chan, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada